CLINICAL TRIAL: NCT04538300
Title: Effect of Chewing Gum on Treatment of Postoperative Nausea-vomiting in Laparoscopic Cholecystectomy: Prospective, Randomized, Controlled Trial
Brief Title: Treatment of Postoperative Nausea-Vomiting in Laparoscopic Cholecystectomy: Peppermint-Flavored Gum Versus Gum-Free
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Canan Yılmaz, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-5/35
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Nausea and Vomiting; Chewing Gum
Keywords: Postoperative Nausea and Vomiting; Chewing gum; Ondansetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: 300 patients ASA I-II, aged between18-65 years who scheduled for elective laparoscopic cholecystectomy under general anesthesia were included. The patients randomly divided into 2 groups (Group G n=150, Group C n=150) with the closed envelope method. In group G peppermint-flavored gum was chewed for 15 minutes in patients with sufficient wakefullness. If PONV persists despite gumming twice, ondansetron iv 4 mg, dexamethasone iv 4 mg, propofol iv 10 mg were given respectively. Patients with moderate and severe nausea in the control group(Group C) were given iv 4 mg ondansetron. If PONV continues, it was planned to give dexamethasone iv 4 mg and propofol iv 10 mg, respectively. In group C(control) degree of nausea and Abramowitz Emezis score were evaluated.
Who Masked: Outcomes Assessor
Masking Description: When efficient wakefullness was gained the participants were asked for nausea and vomiting at recovery room. The outcomes assessor evaluating the participants after the treatment does not know the treatment type made to the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Gum (Active Comparator): Peppermint gum was chewed for 15 minutes in patients with sufficient wakefullness.
  Degree of nausea and Abramowitz Emezis score were evaluated as the interventions. If PONV persists second chewing gum was gived. 15 minutes later PONV was evaluated. If PONV was persisted ondansetron 4 mg, then dexamethasone 4 mg , then propofol 10 mg intravenously were given, respectively.
  Interventions: Diagnostic Test: Abramowitz Emesis Score; Diagnostic Test: Degree of nausea; Diagnostic Test: Observer's Assessment of Alertness/Sedation Scale; Diagnostic Test: Patient Satisfaction; Diagnostic Test: Surgeon Satisfaction; Other: Chewing Peppermint gum
- Group Control (Active Comparator): In Group Control, Degree of nausea and Abramowitz Emezis score were evaluated as the interventions in recovery room. If patients with moderate and severe nausea were given 4 mg ondansetron intravenously. If PONV continues, we planned to give dexamethasone 4 mg and propofol 10 mg intravenously, respectively.
  Interventions: Diagnostic Test: Abramowitz Emesis Score; Diagnostic Test: Degree of nausea; Diagnostic Test: Observer's Assessment of Alertness/Sedation Scale; Diagnostic Test: Patient Satisfaction; Diagnostic Test: Surgeon Satisfaction

INTERVENTIONS:
Diagnostic Test: Abramowitz Emesis Score — Postoperative vomiting was evaluated by Abramowitz emesis score in recovery room.
Diagnostic Test: Degree of nausea — Degree of postoperative nausea was evaluated.
Diagnostic Test: Observer's Assessment of Alertness/Sedation Scale — Patients' sufficient wakefulness was evaluated by Observer's Assessment of Alertness/Sedation scale in the recovery unit.
Diagnostic Test: Patient Satisfaction — Patient satisfaction was questioned. Answers were recorded as one of the choices (never, sometimes, usually or always)
Diagnostic Test: Surgeon Satisfaction — Surgeon satisfaction was questioned. Answers were recorded as one of the choices (never, sometimes, usually or always)
Other: Chewing Peppermint gum — Peppermint gum was chewed for 15 minutes in patients with sufficient wakefullness.
  Arms: Group Gum

SUMMARY:
Postoperative nausea and vomiting (PONV) is an unwanted and distressing complication for patients. PONV affects one-third of untreated patients after general anesthesia. PONV is a hard state for patients, surgeons, and anesthesiologists and increases the anxiety of patient. There are many pharmacologic agents efficient in treatment and prophylaxis of PONV, however, these drugs have many side effects. At the same time, there are many non-pharmacological strategies for antiemetic therapies. Therefore there is an interest to nonpharmacologic agents. Such as acupuncture, ginger, peppermint …etc. Mint is a popular vegetable used as an antispasmodic, analgesic, antimicrobial and anti-vomiting treatment. The use of mint is safe and no certain side-effects and interactions. Chewing affects on postoperative bowel functions. Our hypothesis was mint chewing gum is effective on treatment of PONV. Laparoscopic cholecystectomy surgery has a high risk for PONV in adults. In this study, our aim is to investigate the effect of mint gum chewing in the treatment of PONV in laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
The study protocol was approved by the Local Ethics Committee. Written informed consent was obtained from each patient. The study was carried out in accordance with The Code of Ethics of the Declaration of Helsinki. 300 patients ASA I-II, between18-65 years old, scheduled for elective laparoscopic cholecystectomy under general anesthesia were enrolled in the study. Patients who have pharyngeal or esophageal dysfunction, significant cardiorespiratory dysfunction, phenylketonuria, inadequate to Turkish language comprehension, allergy to mint or antiemetic drugs, were not feasible to chew gum were excluded from the study. All patients were routinely monitored (electrocardiography,SpO2,noninvasive blood pressure). Demographic datas were recorded. Anesthesia induction was made with propofol 2-3mg/kg iv, fentanyl 1.5mcg /kg iv and rocuronium 1mg / kg. Anesthesia maintenance was provided with sevoflurane MAC 1.0 in 50% O2 and air mixture. Intravenous10 mg metoclopromide, 50 mg ranitidine was given to all patients and sugammadex 2 mg/kg were administered for antagonism of neuromusculer block. Before surgical incision paracetamol 1000 mg intravenous was given and 10 minutes before extubation diclofenac sodium 75 mg intramuscular was injected.At the end of surgery the patients were randomly divided into two groups. Group G (Gum group) and Group C (Control group) with the closed envelope method. Patients were followed up in the recovery unit for at least 30 minutes. Degree of nausea and Abramowitz Emezis Score were evaluated for all the patients. In Group G, peppermint gum was chewed for 15 minutes in patients with sufficient wakefulness (Observer's Assessment of Alertness/Sedation scale of 5). The first gum application time was recorded. If patient refused chewing gum, ondansetron iv 4mg was given. If PONV repeated, chewing gum was given again. If PONV was persisted despite chewing gum twice, ondansetron iv 4 mg, then dexamethasone iv 4 mg, propofol 20 mg iv slowly were given, respectively. In Group C, ondansetron 4 mg iv was performed to patients whose postoperative nausea score was bigger than 3 and Abramowitz Emesis score one and above. The first drug application time was recorded. The time of PONV healed fully was recorded. If PONV was continued, it was planned to give ondansetron 4mg iv, dexamethasone 4 mg iv and propofol iv 20 mg iv, respectively. Nevertheless, it was planned to repeat ondansetron 0.15mg / kg at 4-hour intervals in patients whose PONV did not improve, with a total dose not exceeding 16mg. The patients were followed up for 24 hours in terms of PONV. In Group C, sufficient wakefulness was evaluated by Observer's Assessment of Alertness/Sedation scale of 5.If there is a complaint of PONV in the Surgical Service, the gum was given in Group G, then ondansetron 0.15 mg / kg and dexamethasone were given. In Group C,ondansetron 0.15 mg / kg and dexamethasone were given. Additional antiemetic needs, adverse events were recorded postoperatively 24 hours. Patient and surgeon satisfaction were recorded for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* undergone for elective laparoscopic cholecystectomy under general anaesthesia
* American Society of Anesthesiologist (ASA) I-II
* Patients between the ages of 18-65

Exclusion Criteria:

* Patients who did not wish to participate in the study
* Patients who has pharyngeal or oesophagial disfunction
* Significant cardiorespiratory disfunction,
* Phenylketonuria,
* Inadequate to Turkish language comprehension,
* Allergy to mint or antiemetic drugs,
* Patients who was not feasible to chew gum were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Degree of nausea | 24 hours
  Degree of nausea was evaluated as 0=none, 1-3=mild, 4-6=moderate or 7-10=severe. The percentage of patients with mild, moderate or severe nausea were calculated. And also, the percentage of patients without nausea were given.
Emesis | 24 hours
  I used Abramowitz Emesis score. Abramowitz Emesis score was evaluated as 0=No vomiting, 1= slight vomiting (once times), 2=Moderate vomiting (two times), 3= severe vomiting (four times) or 4= Persistent vomiting (continuous).The percentage of patients with sligth, moderate, severe or persistent emesis were calculated. And also, the percentage of patients without emesis were given.

SECONDARY OUTCOMES:
Antiemetic requirement | 24 hours
  Antiemetic drugs were given if nausea score was bigger than 3 and Abramowitz emesis scorewas bigger than 1.
Patient Satisfaction | 24 hours
  Patient satisfaction was questioned. Answers were recorded as one of the choices (0=never, 1=sometimes, 2=usually or 3=always)
Surgeon Satisfaction | 24 hours
  Surgeon satisfaction was questioned. Answers were recorded as one of the choices (0=never, 1=sometimes, 2=usually or 3=always)

CONTACTS AND LOCATIONS:
Overall Officials: Canan Yılmaz, Principal Investigator — Medical Doctor of Anesthesiology Department
Locations (1):
- Bursa Yuksek Ihtisas Education and Research Hospital, Bursa, Turkey (Türkiye)